CLINICAL TRIAL: NCT04081649
Title: Cerebral Oxygenation and Neurological Functioning After Cardiac Surgery
Acronym: CONFUSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Gordon Boyd (Other)
Responsible Party: Sponsor-Investigator, Dr. Gordon Boyd, Associate Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-1672-14
Record Dates: First submitted 2019-06-05; First posted 2019-09-09 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Cognitive Impairment; Delirium
MeSH Terms: conditions — Coronary Artery Disease; Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery: Patients undergoing non-emergent cardiac surgery for coronary bypass graft and/or valvular replacement

SUMMARY:
The overall goal of this research program is to determine quantitative predictors of quantitative long-term neurological functioning following different cardiac surgery procedures. The investigators aim to generate a timeline of neurological function that includes pre-existing performance, post-operative delirium, and neurological outcome. Furthermore, the investigators will test the hypothesis that intraoperative regional cerebral oxygenation (rSO2) desaturations, as measured by near-infrared spectroscopy (NIRS) are associated with poor neurological functioning following cardiac surgery, as measured by a robotic device called the KINARM.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing coronary artery bypass surgery +/- valvular surgery

Exclusion Criteria:

* pre-existing cognitive impairment or neurodegenerative condition
* any reason that participant cannot participate in follow up (lives too far away, limb amputation, speaks language other than english)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing non-emergent surgery will be recruited from the perioperative assessment clinic by a trained researcher.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
12 month cognitive outcome-Repeatable Battery of Neuropsychological Status (RBANS) Total Scale | 12 months
  Participants will be assessed with the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). The RBANS assesses 5 cognitive domains (language, visuospatial, immediate memory, delayed memory, and attention). The individual domain scores are compiled to provide at total cognitive score (Total Scale), which is age-adjusted. The population normative value is 100 +/- 24 (1.96 SD).
12 month cognitive outcome-KINARM robotic assessment-visually guided reaching | 12 months
  This centre-out reaching task assesses basic visuospatial skills and sensorimotor control. The subject's hand is represented by a white dot. Each subject is then instructed to bring the white dot quickly and accurately to the red target as they appear on the screen. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.
12 month cognitive outcome-KINARM robotic assessment-arm position matching | 12 months
  Patients are instructed to mirror-match the movement and final position of the robot-controlled arm. This task is performed twice to obtain data on both arms. Patients will require intact proprioceptive functioning to process information on where their limb is in the horizontal space. This arm position matching task has been shown to determine the degree of position sense impairment in subjects following stroke. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.
12 month cognitive outcome-KINARM robotic assessment-reverse visually guided reaching | 12 months
  This task is presented similarly to the visual guided reaching task. However, the movement of the white dot is now reversed compared to the movement of the patient's hand. To successfully complete the task, patients must move their hand away from the target, thereby reaching the red target with the white dot. This is a more complex reaching task, requiring inhibitory control to not automatically reach towards the red target and a cognitive rule to move the white cursor by moving in the opposite direction. Visuomotor impairments of this nature have been described in individuals at risk of developing Alzheimer's disease. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.
12 month cognitive outcome-KINARM robotic assessment-ball on bar | 12 months
  Patients are instructed to use a virtual bar, generated between their hands, to balance a virtual ball as it appears on the screen. The subject must then bring the balanced ball on bar to different target locations in virtual space. This task consists of three levels: 1) ball fixed to bar, 2) ball moves along bar based on bar orientation, 3) ball can roll freely along bar. This task assesses bimanual motor control. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.
12 month cognitive outcome-KINARM robotic assessment-object hit | 12 months
  In this task, the participants' hands are represented by paddles. Subjects are instructed to hit balls falling down from the top of the screen towards them. As the task progresses, the balls begin to fall more frequently and increase in speed, making the task gradually more difficult. This simple task measures sensorimotor function and decision-making. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.
12 month cognitive outcome-KINARM robotic assessment-object hit and avoid | 12 months
  This task is similar to the object hit task, where patients use the robot's handles to hit objects falling from the top of the screen towards them. In this task however, patients are instructed to only hit two target shapes while avoiding all other shapes (i.e distractors). The Object hit & avoid task therefore requires additional cognitive functions related to attention to identify each shape and inhibitory control to avoid the distractors. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.
12 month cognitive outcome-KINARM robotic assessment-spatial span | 12 months
  A series of squares light up on the screen in a particular sequence. Within a 3-by-4 grid of squares, patients are required to replay the sequence by reaching with their dominant hand to the correct squares. This task assesses visuospatial working memory, and is similar to the Corsi block-tapping task. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.
12 month cognitive outcome-KINARM robotic assessment-trail making | 12 months
  This task is a quantitative version of the standard pen-and-paper neuropsychological test. In trailing making part A, patients are instructed to connect the numbers 1 through 25. The trail making part B task requires subjects to connect the dots by alternating numbers and letters (1-A-2-B-3-C, etc.). This task assesses executive function related to task switching. This task is quantified by several parameters (eg. limb speed, reaction time), which are compiled into an overall task score using the Mahalanobis distance, and further converted to an age-, gender, and handedness matched z-score. A z-score greater than 1.96 is considered abnormal.

SECONDARY OUTCOMES:
Cognitive trajectory (changes in KINARM and RBANS performance from pre-surgery, to 3- and 12-months post-operative) | Pre-operative, 3 months post-operative, and 12-months post-operative
  This will be assessed with the KINARM robot and the RBANS (described above)
Physiological determinants of rSO2 | Intraoperative (3-6 hours)
  Intraoperative hemodynamic and physiological variables will be collected during the operation (eg. mean arterial pressure (mmHg), heart rate (beats per minute), peripheral oxygen saturation (%)) to determine the predictors of rSO2. A linear model will be created to demonstrate the relative contribution each of these predictors has to cerebral oxygenation (rSO2-single outcome variable).

CONTACTS AND LOCATIONS:
Overall Officials: J. Gordon Boyd, MD, PhD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will be willing to share IPD following the publication of our study in peer reviewed literature.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Following publication of our study, our data will be available for 5 years.
Access Criteria: Study PI can be contacted via email for data.

REFERENCES:
- [Derived] Semrau JS, Scott SH, Hamilton AG, Petsikas D, Payne DM, Bisleri G, Saha T, Boyd JG. Road to recovery: a study protocol quantifying neurological outcome in cardiac surgery patients and the role of cerebral oximetry. BMJ Open. 2019 Dec 3;9(12):e032935. doi: 10.1136/bmjopen-2019-032935. PMID 31796491